CLINICAL TRIAL: NCT03978117
Title: Clinical Trial of Two Study Drinks in Detoxification of Environmental Toxicants and Carcinogens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018NTLS144; 2018NTLS144 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze Dried Watercress Preparation (Experimental)
  Interventions: Dietary Supplement: Freeze Dried Watercress Preparation
- Placebo Preparation (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Preparation

INTERVENTIONS:
Dietary Supplement: Freeze Dried Watercress Preparation — Freeze dried watercress containing gluconasturtiin, which when added to provided water with flavor powder, will result in a total target dose of up to 40 mg/day of 2-phenethyl isothiocyanate (PEITC). Preparation consumed at breakfast, lunch and dinner 3x daily for 2 weeks.
  Arms: Freeze Dried Watercress Preparation
Dietary Supplement: Placebo Preparation — Maltodextrin added to provided water with flavor powder. Preparation consumed at breakfast, lunch and dinner 3x daily for 2 weeks.
  Arms: Placebo Preparation

SUMMARY:
The goal of this research is to determine if consuming one of two study drinks will help enhance the detoxification of multiple environmental toxicants and cancer causing agents, particularly in subjects who are null for glutathione-S-transferase M1 (GSTM1), glutathione-S-transferase T1 (GSTT1), or both. If our research supports this idea, this drink could be an inexpensive dietary component, which could promote good health.

DETAILED DESCRIPTION:
Volatile organic carcinogens and toxicants are ubiquitous environmental and endogenous compounds to which virtually all humans are exposed. All of these compounds are detoxified by metabolic processes that ultimately result in conjugation with glutathione and excretion of mercapturic acids in urine. Glutathione conjugation can be upregulated by isothiocyanates through the Nrf2 pathway and related routes of metabolism. This study will examine if watercress consumption, resulting in exposure to milligram amounts of 2-phenethyl isothiocyanate (PEITC) per day, will enhance the detoxification of benzene, acrolein and other related volatile toxicants and carcinogens. One of the two drinks contains PEITC released from freeze dried watercress while the other drink contains maltodextrin.

Benzene causes acute myeloid leukemia/acute non-lymphocytic leukemia in humans, and a positive association has been observed between benzene exposure and acute lymphocytic leukemia, chronic lymphocytic leukemia, multiple myeloma, and non-Hodgkin lymphoma. Acrolein is highly toxic and causes nasal tumors in rats. Benzene is classified as "carcinogenic to humans" by the International Agency for Research on Cancer, and acrolein as "probably carcinogenic to humans." Mercapturic acids of the volatile toxicants and carcinogens propylene oxide, crotonaldehyde, methyl vinyl ketone, methacrolein, and acrylonitrile will also be quantified.

The study will be a randomized, placebo-controlled, single-blind, phase II clinical trial with a crossover study design. Participants will be assigned to active (freeze dried watercress) or placebo (maltodextrin) study product for 14 days, then undergo a 4-week wash-out period, and will then be crossed over to the other product for another 14 days. During the treatment phase, subjects will consume the watercress beverage or placebo, three times per day. The target dose will be 40 mg/day of PEITC. Subjects may be titrated down if they report being unable to tolerate the full dose. Urine, oral swabs, and saliva will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adult Male or female. Participants can be smokers or non-smokers
* In good physical health
* In stable and good mental health
* Not using any medications that may affect the Nrf2 pathway
* Women who are not pregnant or nursing or planning to become pregnant
* Participants have provided written informed consent to participate in the study

Exclusion Criteria:

* Significant immune system disorders, respiratory diseases, kidney or liver diseases or any other medical disorders that may affect biomarker data as determined by the licensed medical professional
* Vital signs outside of the allotted range
* Not willing to abstain from eating cruciferous vegetables during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2024-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PhD, Principal Investigator — University of Minnesota; Stephen Hecht, PhD, Principal Investigator — Department of Laboratory Medicine and Pathology, University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 300 participants randomized to treatment arms. 188 analyzed for study objectives.
Groups:
- Freeze Dried Watercress Preparation Then Placebo: Participants were randomly assigned to the watercress then placebo arm. During the treatment phase, participants consumed the watercress beverage 3 times per day (around the time of breakfast, lunch and dinner) for 14 days. Participants had a 4-week washout period before switching to the placebo beverage for 14 days. The placebo was consumed in the same pattern 3 times per day around meals as the watercress beverage.
- Placebo Then Freeze Dried Watercress Preparation: Participants were randomly assigned to the placebo then watercress arm. During the treatment phase, participants consumed the placebo beverage, 3 times per day (around the time of breakfast, lunch and dinner) for 14 days. Participants had a 4-week washout period before switching to the watercress beverage for 14 days. The watercress beverage was consumed in the same pattern 3 times per day around meals as the placebo beverage.
Period: Overall Study
Arm/Group | Freeze Dried Watercress Preparation Then Placebo | Placebo Then Freeze Dried Watercress Preparation
Started | 155 | 145
Completed | 125 | 115
Not Completed | 30 | 30
Not completed — self- withdrawal or PI withdrawal | 26 | 26
Not completed — Lost to Follow-up | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Freeze Dried Watercress Preparation Then Placebo | Placebo Then Freeze Dried Watercress Preparation | Total
Number analyzed (Participants) | 108 | 80 | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 108 | 80 | 188
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 57 | 126
  Male | 39 | 23 | 62
Race/Ethnicity, Customized [Number; unit: participants]
  Non-White | 25 | 14 | 39
  White | 83 | 66 | 149
Region of Enrollment [Number; unit: participants]
  United States | 108 | 80 | 188

OUTCOME MEASURES:

1. Primary Outcome: Carcinogen Detoxification of Metabolites in Urine.
Description: Carcinogen detoxification metabolites in urine. Biomarkers to be analyzed: 2-cyanoethyl mercapturic acid (CEMA), 3-hydroxypropyl mercapturic acid (HPMA1), 2-hydroxypropyl mercapturic acid (HPMA2), phenyl mercapturic acid (SPMA), 3-hydroxy-1-methylpropyl mercapturic acid (HMPMA1), 3-hydroxy-2-methylpropyl mercapturic acid (HMPMA2), and 3-hydroxy-3-methylpropyl mercapturic acid (HMPMA3),
Time Frame: 2 Months
Population: Number analyzed differs due to incomplete markers in analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Placebo: Maltodextrin added to provided water with flavor powder. Preparation consumed at breakfast, lunch and dinner 3x daily for 2 weeks.
Arm/Group | Freeze Dried Watercress Preparation | Placebo
Number analyzed (Participants) | 188 | 188
ng/mL
  CEMA | 7.26 [4.46 to 19.99] | 6.11 [4.12 to 21.94]
  HPMA1: number analyzed (Participants) | 186 | 187
  HPMA1 | 3052.39 [2249.48 to 5009.80] | 1843.29 [1226.52 to 3395.28]
  HPMA2: number analyzed (Participants) | 188 | 187
  HPMA2 | 329.25 [210.08 to 541.68] | 316.70 [183.33 to 494.16]
  SPMA: number analyzed (Participants) | 188 | 187
  SPMA | 0.60 [0.34 to 1.49] | 0.44 [0.25 to 0.86]
  HMPMA1: number analyzed (Participants) | 180 | 180
  HMPMA1 | 381.91 [281.38 to 507.20] | 307.68 [242.04 to 443.12]
  HMPMA2: number analyzed (Participants) | 183 | 186
  HMPMA2 | 218.68 [161.64 to 335.53] | 180.82 [109.18 to 275.83]
  HMPMA3: number analyzed (Participants) | 169 | 174
  HMPMA3 | 518.58 [441.61 to 646.40] | 388.80 [316.68 to 503.75]
  HMPMA: number analyzed (Participants) | 168 | 175
  HMPMA | 1189.24 [950.12 to 1660.61] | 891.42 [668.65 to 1249.71]

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Freeze Dried Watercress: Freeze dried watercress containing gluconasturtiin, which when added to provided water with flavor powder, will result in a total target dose of up to 40 mg/day of 2-phenethyl isothiocyanate (PEITC). Preparation consumed at breakfast, lunch and dinner 3x daily for 2 weeks.
Arm/Group | Freeze Dried Watercress | Placebo
All-Cause Mortality (participants affected / at risk) | 0/300 | 0/300
Serious Adverse Events (participants affected / at risk) | 0/300 | 0/300
Other Adverse Events (participants affected / at risk) | 188/300 | 50/300
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Freeze Dried Watercress (N=300) | Placebo (N=300)
Saliva, changes in (General disorders) | 1 (1) | 0 (0)
Oral dysesthesia (burning/tingling/numbness/pain) (General disorders) | 21 (21) | 1 (1)
Mouth Sore (General disorders) | 1 (1) | 0 (0)
Dyspepsia (upset stomach) (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastroesophageal Reflux (GERD/heartburn/acid) (Gastrointestinal disorders) | 7 (7) | 3 (3)
Stomach Pain (Gastrointestinal disorders) | 18 (18) | 4 (4)
Vomiting (Gastrointestinal disorders) | 7 (7) | 0 (0)
Nausea (General disorders) | 30 (30) | 5 (5)
Bloating (Gastrointestinal disorders) | 16 (16) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 15 (15) | 3 (3)
Increased gas, belching and changes to stool (Gastrointestinal disorders) | 37 (37) | 8 (10)
Fatigue (General disorders) | 1 (1) | 0 (0)
Vivid Dreams (see S for nightmare/terror) (General disorders) | 1 (1) | 1 (1)
Appetite, Loss of (General disorders) | 4 (4) | 0 (0)
Appetite, Increase/hunger (General disorders) | 1 (1) | 0 (0)
Myalgia (muscle aches/pain/spasms) (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness/Lightheadedness (General disorders) | 2 (2) | 0 (0)
Dysgeusia (change in taste/smell) (General disorders) | 5 (5) | 0 (0)
Headache (incl. migraine) (General disorders) | 4 (4) | 1 (1)
Depressed (sad) mood (Psychiatric disorders) | 1 (1) | 3 (3)
Nightmare/terror (General disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Increased Urination (Gastrointestinal disorders) | 7 (7) | 11 (11)
Nasal congestion (incl. runny nose) (General disorders) | 1 (1) | 0 (0)
Rash (General disorders) | 1 (1) | 0 (0)
Hot Flashes (General disorders) | 1 (1) | 0 (0)
Edema (face/neck/limbs/trunk/localized) (General disorders) | 0 (0) | 1 (1)
Pain (other) (General disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03978117/Prot_SAP_000.pdf
  • Informed Consent Form (2022-09-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03978117/ICF_001.pdf